CLINICAL TRIAL: NCT03904251
Title: A Phase Ib Trial With Dose Expansion Evaluating CPX-351 Plus Gemtuzumab Ozogamicin for Relapsed Acute Myelogenous Leukemia
Brief Title: CPX-351 and Gemtuzumab Ozogamicin in Treating Patients With Relapsed Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Pfizer (Industry); Jazz Pharmaceuticals (Industry); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-001419; NCI-2019-00701 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Acute Myelogenous Leukemia
Keywords: AML, Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Gemtuzumab; CPX-351; Injections; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (CPX-351, gemtuzumab ozogamicin) (Experimental): INDUCTION: Patients receive liposome-encapsulated daunorubicin 44mg/m2 - cytarabine 100mg/m2 IV over 90 minutes on days 1, 3, and 5, and gemtuzumab ozogamicin 3 mg/m2 (max 4.5 mg) IV over 120 minutes on day 7, or days 4 and 7, or days 1, 4, and 7 in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients who achieve CR/CRi receive consolidation therapy at the discretion of the treating physician and/or proceed to allogeneic HSCT.
  Interventions: Drug: Gemtuzumab Ozogamicin; Drug: Liposome-encapsulated Daunorubicin-Cytarabine

INTERVENTIONS:
Drug: Gemtuzumab Ozogamicin — Given IV
  Other Names: Calicheamicin-Conjugated Humanized Anti-CD33 Monoclonal Antibody; CDP-771; CMA-676; gemtuzumab; hP67.6-Calicheamicin; Mylotarg; WAY-CMA-676
Drug: Liposome-encapsulated Daunorubicin-Cytarabine — Given IV
  Other Names: CPX-351; Cytarabine-Daunorubicin Liposome for Injection; Liposomal AraC-Daunorubicin CPX-351; Liposomal Cytarabine-Daunorubicin; Liposome-encapsulated Combination of Daunorubicin and Cytarabine; Vyxeos

SUMMARY:
This phase Ib trial studies the best dose of gemtuzumab ozogamicin when given together with CPX-351 in treating patients with acute myeloid leukemia that has come back after it was previously in remission. CPX-351 is a chemotherapy, which works in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Gemtuzumab ozogamicin is a monoclonal antibody, called gemtuzumab, linked to chemotherapy called calicheamicin. Gemtuzumab attaches to CD33 (transmembrane receptor) positive cancer cells in a targeted way and delivers ozogamicin to kill them. Giving CPX-351 and gemtuzumab ozogamicin may work better in treating patients with acute myeloid leukemia, compared to giving only one of these therapies alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the phase II dose of the combination liposome-encapsulated daunorubicin-cytarabine (CPX-351) plus gemtuzumab ozogamicin (GO) by means of estimating maximum tolerated dose (MTD) in participants with relapsed acute myeloid leukemia (AML).

SECONDARY OBJECTIVES:

I. To estimate the remission rate (complete remission plus complete remission with incomplete hematologic recovery) of participants in the MTD cohort who receive CPX-351 plus GO.

II. To evaluate CPX-351 plus GO as a bridge to allogeneic hematopoietic stem cell transplantation (HSCT) in participants with relapsed AML.

III. To estimate the duration of remission. IV. To evaluate for toxicity by means of Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.

V. To evaluate for the development of veno-occlusive disease at any point during the study in participants treated with CPX-351 plus GO.

VI. To evaluate time to return of normal hematopoiesis after induction therapy. VII. To evaluate 30- and 60-day survival.

EXPLORATORY OBJECTIVES:

I. To evaluate if there is a difference in remission rate based on CD33 splicing single nucleotide polymorphism (SNP) genotype (CC, TC, or TT) in participants receiving CPX-351 plus GO.

II. To evaluate the impact that leukemia cell multidrug resistance activity have on achieving remission after treatment with CPX-351 plus GO.

III. To evaluate the possible associations of participant constitutional genotype, leukemia genotype, and response to therapy.

IV. To evaluate the possible associations of participant ribonucleic acid (RNA) expression, leukemia RNA expression, and response to therapy.

OUTLINE: This is a dose-escalation study of gemtuzumab ozogamicin when given in combination with liposome-encapsulated daunorubicin-cytarabine.

INDUCTION: Patients receive liposome-encapsulated daunorubicin-cytarabine intravenously (IV) over 90 minutes on days 1, 3, and 5, and gemtuzumab ozogamicin IV over 2 hours on day 7 in the first cohort of study participants, days 4 and 7 in the second cohort of study participants, or days 1, 4, and 7 in the third cohort of study participants, in the absence of disease progression or unacceptable toxicity. The dose expansion cohort will receive the above treatment schedule that is determined to be the maximum tolerated dose.

CONSOLIDATION: Patients who achieve complete remission (CR)/CR with incomplete hematologic recovery (CRi) receive consolidation therapy at the discretion of the treating physician and/or proceed to allogeneic HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Bone marrow blasts >= 5% that develops after remission, no restriction on prior number of relapses or regimens
* Eastern Cooperative Oncology Group (ECOG) 0-2
* At least a 3-month duration of remission prior to relapse
* Participants with relapse after allogeneic transplantation are included
* Up to 1 cycle of hypomethylating agent monotherapy at time of relapse is allowed, must be discontinued at least 14 days prior to start of salvage induction
* Serum total bilirubin =< 2.0 mg/dL, unless considered due to Gilbert?s disease or leukemia involvement
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) =< 3 times the upper limit of normal, unless considered due to leukemia involvement
* Alkaline phosphatase =< 3 times the upper limit of normal, unless considered due to leukemia involvement
* Serum creatinine =< 2.0 mg/dL, or creatinine clearance > 40 mL/min based on Cockcroft-Gault glomerular filtration rate (GFR)
* Ability to give full informed consent on their own
* Females of reproductive potential (postmenopausal for less than 24 consecutive months) must have a negative pregnancy

Exclusion Criteria:

* Currently receiving targeted therapy for FLT3 (cytokine receptor tyrosine kinase class III), IDH1, or IDH2 (isocitrate dehydrogenase, 1, 2) mutations and intent to continue use; prior use of targeted therapy for such mutations is allowed, but agents should be discontinued 1 week prior to enrollment
* Acute promyelocytic leukemia
* Second malignancy that would limit survival by less than 2 years
* New York Heart Association class III or VI
* Left ventricular ejection fraction < 50%
* History of coronary stent placement that requires mandatory continuation of dual-antiplatelet therapy
* History of Wilson?s disease or other copper handling disorders
* Hypersensitivity to cytarabine, daunorubicin, or liposomal products
* Active invasive fungal infection
* Active bacterial or viral infection manifesting as fevers or hemodynamic instability within the past 72 hours
* Lifetime cumulative daunorubicin-equivalent anthracycline dose > 368 mg/m^2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to day 42
  MTD is defined as the cohort of participants one cohort below the cohort that develop dose-limiting toxicity (DLT) in at least 2 participants.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to day 42
  Objective response, including complete remission (CR) plus complete remission with incomplete hematologic recovery (CRi), after induction therapy will be measured using the International Working Group (IWG) Response Criteria in acute myeloid leukemia (AML).
Proportion of participants who go on to receive allogeneic hematopoietic cell transplantation (HSCT) after achieving CR/CRi | Up to 18 months
  The proportion of patients who receive an allogeneic HSCT following a CR/CRi response will be reported along with an exact 95% confidence interval.
Duration of remission | Up to 18 months
  Evaluated in participants that achieve CR/CRi, and defined as number of days that elapse from first day CR/CRi to the first day that bone marrow blasts >= 5%. The median duration of remission will be reported in patients who achieved CR/CRi, along with the corresponding range.
Incidence of toxicities | Up to day 42
  Measured by the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Diagnosis of veno-occlusive disease (VOD) | Up to 18 months
  The diagnosis of veno-occlusive disease is based on the Baltimore criteria: Bilirubin > 2.0 mg/dL, plus, painful hepatomegaly, ascites, and weight gain > 5% basal since initiating therapy with gemtuzumab ozogamicin (GO). The proportion of patients who develop VOD will be reported along with an exact 95% confidence interval.
Time to return of normal hematopoiesis | From day 1 of induction, assessed up to 18 months
  Defined as the number of days from day 1 of induction to ANC (absolute neutrophil count) >= 1000/uL (upper limit) and platelet count >= 100,000/uL. Will be reported along with the corresponding range.
Number of participants deceased at day 30 and day 60 | At 30 and 60 days following the start of induction
  Mortality is defined as death having occurred in any participant that receives at least one dose of experimental therapy. Kaplan-Meier methods will estimate the overall survival at day 30 and day 60 following the start of induction. The survival estimate at these two time points will be reported along with a 95% confidence interval.

OTHER OUTCOMES:
Genotype at CD33 splicing single nucleotide polymorphism (SNP) RS12459419 | Up to 18 months
  Determined by whole exome sequencing and confirmatory genotyping.
Multidrug resistance activity of leukemia cell P-glycoprotein (Pgp) | Up to 18 months
  Will be determined by the flow cytometry mean fluorescence intensity (MFI) of the efflux of the fluorescent dye DiOC2 (Diethyloxacarbocyanine iodide) (by malignant cells. Will be assessed by dye efflux assay as described by Walter et al. 2003.
Multidrug resistance activity of leukemia cell multidrug resistance protein 1 (MRD1) | Up to 18 months
  Will be determined by the flow cytometry efflux MFI of the efflux of the fluorescent dye 5-carboxy-2?,7?-dichlorofluorescein diacetate (CDCF) by malignant cells. Will be assessed by dye efflux assay as described by Walter et al. 2003.
Exome sequencing analysis | Up to 18 months
  Tumor deoxyribonucleic acid (DNA) and participant DNA will be measured via Illumina HiSeq3000 sequencing platform to evaluate for associations between participant constitutional genotype (buccal swab sample at enrollment), leukemia genotype (bone marrow aspirate at enrollment and upon relapse), and response to therapy.
Ribonucleic acid (RNA) sequencing analysis | Up to 18 months
  Tumor RNA and participant RNA will be measured via RNA sequencing technique.

CONTACTS AND LOCATIONS:
Overall Officials: Caspian Oliai, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (5):
- United States (5):
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of California San Diego, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California

REFERENCES:
- [Derived] Jentzsch M, Grimm J, Bill M, Brauer D, Backhaus D, Goldmann K, Schulz J, Niederwieser D, Platzbecker U, Schwind S. ELN risk stratification and outcomes in secondary and therapy-related AML patients consolidated with allogeneic stem cell transplantation. Bone Marrow Transplant. 2021 Apr;56(4):936-945. doi: 10.1038/s41409-020-01129-1. Epub 2020 Nov 19. PMID 33208914